CLINICAL TRIAL: NCT04312347
Title: Tamoxifen Dose Adjustment on ER+ Breast Cancer Patients Based on Genomic and Metabolite Concentrations Analysis
Brief Title: Tamoxifen Dose Adjustment on Indonesian Female ER+ Breast Cancer Patients Based on CYP2D6 Genotype and Endoxifen Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nalagenetics Pte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMS01190510
Record Dates: First submitted 2020-03-05; First posted 2020-03-18 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2020-03

CONDITIONS: ER+ Breast Cancer
Keywords: breast cancer; tamoxifen; CYP2D6; endoxifen
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized dosing of tamoxifen (Experimental): Increase tamoxifen dose into 40 mg/day for patients with low endoxifen level and poor/intermediate metabolizer CYP2D6 phenotype.
  Interventions: Drug: Tamoxifen dose adjustment

INTERVENTIONS:
Drug: Tamoxifen dose adjustment — Patients with low endoxifen level and poor/intermediate metabolizer CYP2D6 phenotype will receive tamoxifen dose escalation into 40 mg/day.

SUMMARY:
The objectives of this study is to perform CYP2D6 genotyping and metabolite concentrations analysis on ER+ breast cancer patients who are taking tamoxifen and give dose recommendations based on the CYP2D6 genotypes and endoxifen levels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ER+ breast cancer
* Have taken tamoxifen daily for at least 2 months

Exclusion Criteria:

* Have not taken tamoxifen daily for at least 2 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Effects of genotype and phenotype of CYP2D6 on plasma and serum concentration of tamoxifen and its metabolites | 8 weeks after initial tamoxifen intake
Effects of dose recommendation of tamoxifen based on CYP2D6 genotyping results on endoxifen levels | 8 weeks after dose recommendation
Frequencies of CYP2D6 alleles in female Indonesian population | Baseline, pre-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Baitha P. Maggadani, Principal Investigator — Department of Pharmacy, University of Indonesia
Locations (1):
- MRCCC Siloam Hospital Semanggi, Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Madlensky L, Natarajan L, Tchu S, Pu M, Mortimer J, Flatt SW, Nikoloff DM, Hillman G, Fontecha MR, Lawrence HJ, Parker BA, Wu AH, Pierce JP. Tamoxifen metabolite concentrations, CYP2D6 genotype, and breast cancer outcomes. Clin Pharmacol Ther. 2011 May;89(5):718-25. doi: 10.1038/clpt.2011.32. Epub 2011 Mar 23. PMID 21430657
- [Background] Fox P, Balleine RL, Lee C, Gao B, Balakrishnar B, Menzies AM, Yeap SH, Ali SS, Gebski V, Provan P, Coulter S, Liddle C, Hui R, Kefford R, Lynch J, Wong M, Wilcken N, Gurney H. Dose Escalation of Tamoxifen in Patients with Low Endoxifen Level: Evidence for Therapeutic Drug Monitoring-The TADE Study. Clin Cancer Res. 2016 Jul 1;22(13):3164-71. doi: 10.1158/1078-0432.CCR-15-1470. Epub 2016 Feb 4. PMID 26847054